CLINICAL TRIAL: NCT05164419
Title: Impact de la Marge de résection Sur la Survie à Long Terme et le Taux de récidive Des Patients Atteints de Cancers Colorectaux opérés au CHUS Entre 2006 et 2016 Pour Des métastases hépatiques
Status: Completed | Type: Observational
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-1611
Record Dates: First submitted 2021-12-07; First posted 2021-12-20 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Colorectal Cancer Stage IV
Keywords: liver surgery; Colorectal liver metastasis
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Wide margin: Patients who underwent surgery with a final pathologic margin of more than 5mm.
- Close margin: Patients who underwent surgery with a final pathologic margin of less than 5mm

SUMMARY:
We retrospectively looks at the impact of the margin status and its size in mm on the recurrence rate in colo-rectal liver metastasis surgery.

DETAILED DESCRIPTION:
Main objective : evaluation the margin status (<1mm, 1-4mm, 5-9mm, >10mm) on the survival and recurrence in colo-rectal liver metastases surgery.

Secondary objectives include :

Evaluate potentiel effects of neo-adjuvant chemotherapy, portal embolisation, and evaluate potentiel bias such as size and number of liver metastases, TNM status of original tumor, timing between primary and metastasis, and extra-hepatic disease.

Methods :

A retrospective cohort study is built where all patients undergoing liver surgery for colorectal liver metastases between 2011 and 2015 are analysed. Subjects are separated in groups according to their margin status. The local and distal recurrence rates are measured and well as survival. Data is obtained through our hospital data management system. Inclusion criterias include age over 18, primary colorectal cancer metastatic to the liver, having undergone surgery between 2011 and 2015, available pathology reports with required data, available radiologic follow-up. Exclusion criterias include repeat liver resection, documented grossly positive margins (R2 resection), and unavailable pathologic information and follow-up. Using survival as primary outcome (Kaplan Meier) and considering 25% potential loss to follow-up, we calculated a sample size. Since this a retrospective study, no patient is directly contacted. Data will is handled by the surgery resident responsible for the project as well as by research assistants. Statistical analysis are performed accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Primary colorectal cancer with liver metastasis
* Undergone liver surgery at our center between 2011 and 2015
* Pathological reports with margin status available (or specimen still available for measurement)

Exclusion Criteria:

* Repeat liver resection No tissu or incomplete pathological information

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with colorectal liver metastases undergoing liver resection at our institution during the defined time-frame.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2006-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Overall survival | 2 years
  Patient is dead or aline

SECONDARY OUTCOMES:
Local recurrence | 2 years
  Advent of recurrence in the liver parenchyma, measured by any time of medical imaging
Distant recurrence | 2 years
  Advent of recurrence anywhere other than liver, measured by any time of medical imaging